CLINICAL TRIAL: NCT05103592
Title: Assessment of Tartrate- Resistant Acid Posphatase 5b (TRACP-5b) in Primary and Secondary Osteoprosis
Brief Title: Assessment of TRACP-5b in Primary and Secondary Osteoporosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Mohammad Abdalmageed Mansour, resident doctor at Rheumatology and Rehabilitation department, Assiut University
Other Study IDs: TRACP-5b in Osteoprosis
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Osteoporosis
Keywords: primary and secondary
MeSH Terms: conditions — Osteoporosis; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Primary osteoprosis patients: patients older than 18 years with primary osteoporosis diagnosed by dxa scan . tartrate- resistant acid phosphatase 5b level will be measured.
  Interventions: Diagnostic Test: Tartrate- resistant Acid Phosphatase marker
- Rheumatoid arthritis patients: patients older than 18 years with primary osteoporosis diagnosed by dxa scan and rhumatoid arthritis.
  tartrate- resistant acid phosphatase 5b level will be measured.
  Interventions: Diagnostic Test: Tartrate- resistant Acid Phosphatase marker
- Ankylosing spondylitis patients: patients older than 18 years with primary osteoporosis diagnosed by dxa scan and ankylosing spondylitis.
  tartrate- resistant acid phosphatase 5b level will be measured.
  Interventions: Diagnostic Test: Tartrate- resistant Acid Phosphatase marker
- Control group: patients older than 18 years not complaining of any bone disease tartrate- resistant acid phosphatase 5b level will be measured.
  Interventions: Diagnostic Test: Tartrate- resistant Acid Phosphatase marker

INTERVENTIONS:
Diagnostic Test: Tartrate- resistant Acid Phosphatase marker — marker could be diagnostic for osteoporosis

SUMMARY:
Assessment of the TRACP-5b level in 1ry OP and 2ry OP such as RA and seronegative spondylitis, that may help in surrogating the use of BMD.

DETAILED DESCRIPTION:
Osteoporosis is a disease characterized by low bone density and a deterioration of bone microarchitecture that reduces bone strength and increases the risk of fracture. The hallmark of osteoporosis is the loss of both bone mineral and bone matrix. Although Bone mass density (BMD) is still the gold standard for the diagnosis of osteoporosis, but bone turnover markers (BTMs) can provide helpful information regarding the bone remodelling process. One of these relatively recent markers is the Tartrate-resistant acid phosphatase (TRACP). TRACP, which was first identified in human leukocytes, has 2 isoforms TRAP-5a derived from macrophages and dendritic cells and TRACP-5b secreted by osteoclasts. it is believed that TRACP-5b is a useful marker of osteoclast activity, even a marker for osteoclast number, as it is associated with osteoclast differentiation, activation and proliferation. Furthermore, it has the advantage of not being affected by renal dysfunction, nor food intake and has a weak diurnal variability. And this is why it has been used as one of the bone turnover markers in evaluating the efficacy of different anti-resorptive treatments in postmenopausal osteoporosis and in 2ry OP due to rheumatoid arthritis as well as in evaluating its specificity in identification of postmenopausal OP when compared to measurement of more expensive, relatively unavailable bone mineral density (BMD).So far, limited researches are available regarding the TRACP-5b level difference among 1ry OP (postmenopausal women) and 2ry OP (ex. RA, SpA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with 1ry OP diagnosed by DXA scan .
* Any RA and SpA patients (older than 18 years old), who fulfill the for mentioned diseases criteria with secondary osteoporosis as diagnosed by DXA scan.

Exclusion Criteria:

* Patients unwilling to participate in the study.
* Patients with other autoimmune diseases.
* Patients depending on Glucocorticoids with in the last 6 month.
* Patients with other causes of 2ry OP (ex. Endocrinal abnormalities, Gastrointestinal diseases, Renal diseases…..etc.)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult 1ry osteoporotic, rheumatoid arthritis and seronegative spondylitis patients who consecutively attend the inpatient unit or outpatient clinic of Rheumatology, Rehabilitation and Physical Medicine Department, Assiut University Hospitals will be recruited in the study.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the TRACP-5b level in 1ry OP and 2ry OP such as RA and seronegative, that may help in surrogating the use of BMD. | Baseline
  Assessing Tartrate- resistant Acid Phosphatase Marker in primary osteoporosis, rheumatoid arthritis, ankylosing spondylitis and control group that may help in substituting Dxa scan.

CONTACTS AND LOCATIONS:
Overall Officials: AMIRA MA MANSOUR, Principal Investigator

REFERENCES:
- [Background] Mederle OA, Balas M, Ioanoviciu SD, Gurban CV, Tudor A, Borza C. Correlations between bone turnover markers, serum magnesium and bone mass density in postmenopausal osteoporosis. Clin Interv Aging. 2018 Aug 3;13:1383-1389. doi: 10.2147/CIA.S170111. eCollection 2018. PMID 30122910
- [Background] Assessment of fracture risk and its application to screening for postmenopausal osteoporosis. Report of a WHO Study Group. World Health Organ Tech Rep Ser. 1994;843:1-129. No abstract available. PMID 7941614
- [Background] Tahtela R, Seppanen J, Laitinen K, Katajamaki A, Risteli J, Valimaki MJ. Serum tartrate-resistant acid phosphatase 5b in monitoring bisphosphonate treatment with clodronate: a comparison with urinary N-terminal telopeptide of type I collagen and serum type I procollagen amino-terminal propeptide. Osteoporos Int. 2005 Sep;16(9):1109-16. doi: 10.1007/s00198-004-1819-7. Epub 2004 Dec 17. PMID 15605190
- [Background] Mochizuki T, Yano K, Ikari K, Okazaki K. Effects of romosozumab or denosumab treatment on the bone mineral density and disease activity for 6 months in patients with rheumatoid arthritis with severe osteoporosis: An open-label, randomized, pilot study. Osteoporos Sarcopenia. 2021 Sep;7(3):110-114. doi: 10.1016/j.afos.2021.08.001. Epub 2021 Aug 27. PMID 34632114